CLINICAL TRIAL: NCT06423625
Title: Developing a Prediction Score Model for Predicting the Likelihood of Hemorrhagic MI Before Percutaneous Coronary Reperfusion Therapy
Brief Title: Hemorrhagic MI Prediction Score Model
Acronym: MIRON-PRE-xAI
Status: Completed | Type: Observational
Sponsor: Rohan Dharmakumar (Other)
Responsible Party: Sponsor-Investigator, Rohan Dharmakumar, Executive Director, Krannert Cardiovascular Research Center, Indiana University School of Medicine
Organization: Indiana University (Other)
Other Study IDs: 19978d
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; Prediction Score; Machine Learning; Hemorrhagic MI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Developing a prediction score model for predicting the likelihood of Hemorrhagic MI

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yrs
* Index MI
* Primary PCI

Exclusion Criteria:

* History of prior myocardial infarction,
* Thrombolysis before PCI
* Contraindication to Cardiac MRI

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of individuals aged 18 - 80 yrs who have been diagnosed with acute ST-elevation myocardial infarction (STEMI) and are scheduled for emergency percutaneous coronary intervention (PCI).
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
Hemorrhagic MI | Emergency admission to Percutaneous Intervention
  Percentage of MI patients confirmed as Hemorrhagic MI

CONTACTS AND LOCATIONS:
Overall Officials: Keyur P Vora, MD FACC, Principal Investigator — Indiana University School of Medicine, Krannert Cardiovascular Research Center
Locations (1):
- Krannert Cardiovascular Research Center, Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No